CLINICAL TRIAL: NCT06922487
Title: Förekomsten av trötthet Vid Neurokirurgisk Vakenkirurgi
Brief Title: Assessment of Tiredness During Awake Resection of Intracerebral Tumors
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01935-01 study 4
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Brain Tumor Adult; Awake Surgery
Keywords: open resection of intracranial tumor; awake surgery; sleepiness
MeSH Terms: conditions — Sleepiness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- awake surgery: intracranial tumor resection via awake surgery, adult.
  Interventions: Procedure: Karolinska Sleepiness Scale, KSS

INTERVENTIONS:
Procedure: Karolinska Sleepiness Scale, KSS — Assessment of sleepiness during resection using KSS

SUMMARY:
Occasional patients with intracranial tumors need to have a planned awakening during surgery to avoid major disability from the tumor resection. During the awake part of the surgery an increasing degree of tiredness is observed. For the surgeon to plan the resection knowledge of the degree and speed of tiredness/sleepiness evolution is important.

The goal of this single center study is to use the "Karolinska Sleepiness Scale" during and after awake surgery for neurosurgical tumor resection to quantify the time available for surgical intervention.

Participants are adults having planned surgery for open resection of intracranial tumor with a planned awakening for assessment during surgery. Participants will be asked to grade postoperative sleepiness using the "Karolinska Sleepiness Scale".

DETAILED DESCRIPTION:
Background The incidence of primary tumors in the central nervous system in adults in Sweden is approximately 1400 per year. Gliomas constitutes the most common form, approximately 50%. The neurosurgery aims at securing material for pathological-anatomical diagnosis, reduction of symptoms, maximal reduction of tumor mass with minimal functional impact. Occasional patients present with tumors in sensitive areas necessitating operation with the patient awake and co-operable to optimize the resection. The procedure is typically performed as an asleep-awake-asleep procedure. A clinical observation is that the patients tend to become increasingly sleepy/tired during resection. This study aims to quantify this phenomenon.

Methods Ethical review board approval (Dnr 2024-01935-01, Stockholm, Sweden) is present.

The study is a single center kohort study.

Participants will be identified by the neurosurgeon planning tumor resection with intraoperative awake surgery. Inclusion and information are given preoperatively by the neurosurgeon and the anesthetist.

All participants receive propofol/remifentanil based general anesthesia with norepinephrine infusion to support blood-pressure during preparation and craniotomy whereafter the participant is awakened. The resection starts when the participant is coherent and cooperative. Peroperative level of sedation is assessed using Karolinska Sleepiness Scale (KSS) every 15 minutes. KSS is an ordinal nine grade scale assessing sleepiness during the last five minutes from "extremely alert" to "very sleepy, great effort to keep awake, fighting sleep". When the resection is completed the participants receives general anesthesia during wound closure. Postoperative level of sedation is assessed using Karolinska Sleepiness Scale (KSS) during the first two postoperative hours.

Data regarding age, sex, length, weight, comorbidities, tumor location, ASA- classification and preoperative medication will be collected. Peroperative vital parameters and pEEG -results and data from infusion pumps are primarily collected electronically. The manually kept anesthetic notes are copied and stored as back-up. All individual data are de-identified and coded after collection.

Inclusion and exclusion criteria Inclusion Adult (>18 years old) Elective supra or infratentorial tumor resection via craniotomy Surgical need for awake surgery Cognitive function allowing informed consent.

Exclusion Tumor localization not allowing placement of BIS electrodes due to interference with surgery Morbid obesitas

Outcomes Peroperative degree of sleepiness measured with Karolinska Sleepiness Scale (KSS).

Statistical methods and power calculation The study is a descriptive cohort study. A convenience sample of participants fulfilling inclusion criteria during the inclusion time will be used. The primary goal is to include at least 10 participants. As primary KSS variable a deviation of two or more units will be considered a significant change. Time from start of resection until significant change in KSS is the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old)
* Elective supra or infratentorial tumor resection via craniotomy
* Surgical need for awake surgery
* Cognitive function allowing informed consent.

Exclusion Criteria:

* Tumor resection without awake surgery
* Morbid obesitas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants presenting to the neurosurgical unit, Skane University hospital, Lund, Sweden for resection of intracranial tumor via craniotomy assessed to benefit from awake surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in KSS | during surgery and 2 hours postoperatively
  Change in KSS during resection

CONTACTS AND LOCATIONS:
Overall Officials: Malin Rundgren, MD, PhD, Principal Investigator — Anaesthesia and Intensive Care, Skane University hospital, Lund, Sweden
Locations (1):
- Intensive and Perioperative Care, Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
IPD will probably be shared after publication.